CLINICAL TRIAL: NCT05065905
Title: A I//II Phase Study of the Efficacy and Safety of Interferon-Gamma by Subcutaneous Injection in the Complex Treatment of Patients Infected With HIV and Tuberculosis
Brief Title: Study of Interferon-Gamma in the Complex Treatment of Patients Infected With HIV and Tuberculosis
Acronym: MSPB_TB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SPP Pharmaclon Ltd. (Industry)
Collaborators: North-Western State Medical University named after I.I.Mechnikov (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSPB_TB
Record Dates: First submitted 2021-09-07; First posted 2021-10-04 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2021-09

CONDITIONS: HIV Coinfection; Aids/Hiv Problem; Tuberculosis, Pulmonary; Human Immunodeficiency Virus; Lentivirus Infections; RNA Virus Infections
Keywords: interferon gamma, IFN-g, HIV infection, tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis, Pulmonary; Acquired Immunodeficiency Syndrome; Lentivirus Infections; RNA Virus Infections; Tuberculosis | interventions — Interferon-gamma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interferon (Experimental): All participants receive subcutaneous interferon-gamma (Ingaron®) 500,000 IU alternated with Interal® (interferon alpha) 3,000,000 IU every other day
  Interventions:
  Drug: Ingaron® Drug: Interal® Drug: Antituberculosis complex therapy
  Interventions: Drug: Interferon-Gamma
- Interferon daily (Experimental): All participants receive subcutaneous interferon-gamma (Ingaron®) 500,000 IU given with Interal® (interferon alpha) 3,000,000 IU every day
  Interventions:
  Drug: Ingaron® Drug: Interal® Drug: Antituberculosis complex therapy
  Interventions: Drug: Interferon-Gamma
- Control (No Intervention): All participants receive only basic antimicrobial treatment
  Interventions:
  Drug: Antituberculosis complex therapy

INTERVENTIONS:
Drug: Interferon-Gamma — received by microbiological synthesis; specific antiviral activity on cells is 2x10*7 Units per mg of protein
  Other Names: Ingaron; Interferon gamma human recombinant
  Arms: Interferon; Interferon daily

SUMMARY:
The primary purpose of this study is to assess the safety and efficacy of interferon-gamma by subcutaneous injection in complex treatment of patients with co-infection of HIV and pulmonary tuberculosis and to determine the rational of its use.

DETAILED DESCRIPTION:
Study will evaluate safety and efficacy of the investigational medical product (IMP) - interferon-gamma - in participants with HIV-infection and pulmonary tuberculosis.

Interferon-gamma (immune interferon) is an important anti-inflammatory cytokine produced by NK-cells, CD4 Th1 cells and CD8 cytotoxic supressor cells. Interferon-gamma blocks viral replication, viral proteins synthesis and assembly of mature viral particles. Causes cytotoxic effects on the cells infected by intracellular pathogens. Possess a bright immunomoduling action. Thus, the use of interferon-gamma is patogenetically rational in patients co-infected with tuberculosis and HIV.

The aim of interferon-gamma use is to achieve a viral replication control, support CD4 level and help abacillation process. In this randomised, controlled safety and efficacy study interferon gamma will be administered in a daily dose of 500,000 IU daily or every other day.

The treatment regimen in this study will also include a basic antituberculosis therapy.

The available clinical data do not suggest a risk for serious adverse events (SAEs) from the IMP used in chosen doses.

The study will screen HIV-infected participants 18-50 years old with pulmonary tuberculosis. Participants who provide informed consent and meet study entry criteria will be randomised into 1 of 3 parallel treatment groups. The study will last 30 days, during which participants will receive IMP in various regimens according to the group.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign the form of informed consent and agree to follow the protocol requirements
* Women willing to participate in the study must protect against possible pregnancy during all the study long
* Age 18-50 years
* Pulmonary tuberculosis
* HIV/AIDS
* Indication for in-patient standard antituberculosis treatment

Exclusion Criteria:

* Investigational research agents received within 30 days before the screening and participation in other clinical trials
* Immunosuppressive medications received within 6 months before the screening
* Current drug abuse for more than 3 years
* Contraindications to interferons of standard antimicrobial therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2006-01-19 (Actual); Primary Completion 2006-03-29 (Actual); Study Completion 2006-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Shmelev, Doctor, Study Director — SPP Pharmaclon Ltd.
Locations (2):
- Russia (2):
  - Saint-Petersburg State Medical Academy n.a. I.I.Mechnikov of Ministry of Health, Saint Petersburg, Sankt-Peterburg
  - City Tuberculosis Hospital #2 of Saint-Petersburg, Saint Petersburg, Sankt-Peterburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon: All participants receive subcutaneous interferon-gamma (Ingaron®) 500,000 IU alternated with Interal® (interferon alpha) 3,000,000 IU every other day
  Interventions:
  Drug: Ingaron® Drug: Interal® Drug: Antituberculosis complex therapy
  Interferon-Gamma: received by microbiological synthesis; specific antiviral activity on cells is 2x10*7 Units per mg of protein
- Interferon Daily: All participants receive subcutaneous interferon-gamma (Ingaron®) 500,000 IU given with Interal® (interferon alpha) 3,000,000 IU every day
  Interventions:
  Drug: Ingaron® Drug: Interal® Drug: Antituberculosis complex therapy
  Interferon-Gamma: received by microbiological synthesis; specific antiviral activity on cells is 2x10*7 Units per mg of protein
Period: Overall Study
Arm/Group | Interferon | Interferon Daily | Control
Started | 30 | 28 | 20
Completed | 30 | 28 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interferon | Interferon Daily | Control | Total
Number analyzed (Participants) | 30 | 28 | 20 | 78
Age, Customized [Count of Participants; unit: Participants]
  under 18 y.o. | 0 | 0 | 0 | 0
  18-50 y.o. | 30 | 28 | 20 | 78
  over 50 y.o. | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 30 | 28 | 20 | 78
Region of Enrollment [Number; unit: participants]
  Russia | 30 | 28 | 20 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sputum Culture
Description: Precentage of participants with negative sputum culture
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Interferon | Interferon Daily | Control
Number analyzed (Participants) | 30 | 28 | 20
Participants | 15 | 20 | 14

2. Secondary Outcome: Average Hemoglobin Level
Description: Level of hemoglobin (g/L)
Time Frame: Screening, Week 8
Reporting Status: Not Posted

3. Secondary Outcome: Leucocytes Level
Description: Number of leukocytes
Time Frame: Screening, Week 4
Reporting Status: Not Posted

4. Secondary Outcome: CD3
Description: CD3 cells level in absolute numbers and percents
Time Frame: Screening, Week 4
Reporting Status: Not Posted

5. Secondary Outcome: CD4
Description: CD4 cells level in absolute numbers and percents
Time Frame: Screening, Week 4
Reporting Status: Not Posted

6. Secondary Outcome: CD8
Description: CD8 cells level in absolute numbers and percents
Time Frame: Screening, Week 4
Reporting Status: Not Posted

7. Secondary Outcome: CD4/CD8
Description: Immunoregulatory index value
Time Frame: Screening, Week 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Interferon | Interferon Daily | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/20
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No